CLINICAL TRIAL: NCT06716450
Title: A Study to Evaluate the Accuracy, Usability and Readability of the Multiplo® TP/HIV Antibody Self-Test Performed by Observed Intended Users in Canada and the Impact of Peer-led HIV and Syphilis Care Among People Experiencing Homelessness in Toronto
Brief Title: Multiplo Tp/HIV Self-Test
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: REACH Multiplo ST-01
Record Dates: First submitted 2024-11-18; First posted 2024-12-04 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: HIV Infection; Syphilis Infection
Keywords: self-test; device trial; screen test
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Screening for HIV and syphilis infection at point of care settings as a self-test in the presence of a trained, silent observer. The embedded study will involve participants interacting with a peer navigator following the self-test to discuss prevention and care options for HIV and syphilis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with unknown HIV and syphilis status (Experimental): All participants will self-test fingerstick blood testing with the test device, along with venous blood testing at a central laboratory using licensed gold standard comparator methods.
  Interventions: Device: Multiplo TP/HIV Antibody Test

INTERVENTIONS:
Device: Multiplo TP/HIV Antibody Test — The Multiplo TP/HIV Antibody Test (MedMira Laboratories Inc., Halifax, NS), ["Multiplo TP/HIV Test"] is a single use, rapid, vertical-flow in vitro qualitative immunoassay for the detection of antibodies to Human Immunodeficiency Virus (HIV) Type 1/Type 2 and Treponema pallidum (Syphilis) in human fingerstick blood. The Multiplo® TP/HIV Test is intended as an aid in the diagnosis of HIV1/2 and Syphilis infections in patients with signs and symptoms of HIV and syphilis. The test is intended for use by trained personnel in medical facilities, clinical laboratories, emergency care situations, and physicians' offices as an in vitro diagnostic device capable of providing results in less than five minutes. The Multiplo TP/HIV Test has not yet sought approval for self-testing. All required pre and post-test counselling guidelines must be followed in each setting in which the Multiplo TP/HIV Test is used. Results are read visually.

SUMMARY:
To help reach the undiagnosed living with HIV and/or syphilis in Canada, self-tests for HIV and Syphilis may have substantial utility for increased identification of infected individuals through their relative ease of use and portability, as well as their ability to deliver rapid, actionable results while the care provider still has access to the patient. MedMira Laboratories Inc. (Halifax, Nova Scotia, Canada) has developed a point-of-care (POC) test to detect HIV and Syphilis antibodies in fingerstick blood samples that is under final review by Health Canada for use by trained Healthcare professionals. A self-test version of this test, with simplified instructions for use has been developed for investigational studies. The goal of the following study sponsored by REACH Nexus is to provide evidence that untrained lay persons / intended users can perform the Multiplo Tp/HIV Self-Test without any increased risk of obtaining erroneous results.

DETAILED DESCRIPTION:
This is a cross-sectional study that employs both observational and interview-based methods. All participants will read the instructions for use (IFU) and conduct the Multiplo TP/HIV Self-Test. They will not be provided any training prior to use. A trained Observer will observe and document the use of the test and independently read the lay user self-test result. 400 participants will also be provided with ten (10) mock devices with different results and asked to interpret those results (i.e. strong positive, weak positive, negative, invalid with no control line and no test dots, and invalid with no control line and positive test dots). The participants will then complete a questionnaire to share their opinions on usability and label comprehension of this test.

All participants will also have a venous blood sample collected for testing of serum at a central laboratory with a 4th generation HIV EIA and standard syphilis serology that will serve as the Comparator Methods (CM). All self-tests will be confirmed using laboratory-standard HIV and syphilis testing algorithms. The sensitivity and specificity of the self-test results will be calculated relative to the "clinical truth" of the participants' HIV and syphilis status determined by the comparator methods.

All enrolled Participants will voluntarily provide medical history and the specimens according to Section 4, Study Procedures at Visit 1 (Day 1), for the testing with the Multiplo TP/HIV Self-Test. Persons with reactive syphilis self-tests may be counselled for immediate treatment.

All Participants will have a laboratory test done for performance comparison and will be instructed to return to the clinic for a follow-up visit (Visit 2), two (2) weeks later to obtain their laboratory test results. Participants may also have a separate Point-of-Care (POC) test for HIV and/or syphilis conducted on-site as part of the clinic's standard of care testing, outside of the protocol.

* Subject recruitment
* Registration and confirmation of eligibility (enrolment questionnaire)
* Administering informed consent
* Review of inclusion/exclusion criteria and enrollment
* Venous blood specimen collection for laboratory testing
* Participant brought to a private room with site observer
* Observer instructs participant on study process (not testing procedure)
* Participant given one Multiplo Tp/HIV Self-Test package
* Participant performs the self-test and interprets the results
* Observer then interprets the participant's self test results
* Observer interviews participant with self-test questionnaire
* Participant given the option of participating in the Mock Result Interpretation exercise
* Participant returns to the site for the laboratory results in approximately 2 weeks

MOCK RESULTS INTERPRETATION A minimum of 400 participants across all study sites will complete device interpretation of contrived (mock) results from prepared devices. Devices will include contrived reactive, weakly reactive, negative, and 2 types of invalid results with their reactivity blinded to the participant.

ELIGIBILITY:
Inclusion Criteria:

* Are ≥18 years of age.
* Can speak/read/write English or French.
* Have presented for voluntary testing for HIV and/or syphilis infection in the clinic or community-based setting.
* Are willing to participate in the study site's standard of care HIV and syphilis counselling and testing program and receive the study site's standard of care test results.
* Are willing to be a participant in the study.
* Can provide informed consent i.e. understand and sign or instruct the Observer to sign the informed consent form.
* Can complete the required testing on the allocated testing day.
* Are willing to provide the necessary fingerstick and venipuncture blood for use in the study protocol testing methods.
* Are of unknown HIV and syphilis status (last HIV and syphilis negative test must be a minimum of 3 months prior).

Exclusion Criteria:

* Do not meet the inclusion criteria.
* Are known HIV and/or syphilis positive.
* Have ever tested positive for syphilis or HIV at any time.
* Have any experience in conducting rapid point-of-care tests on patients for HIV, syphilis or any other infectious disease.
* Are familiar with the Multiplo® TP/HIV Self-Test.
* Are investigator site employees or immediate family members of sponsor or investigator sites.
* Have participated in any prior, or concurrent trial of HIV and syphilis self-tests.
* Are a practicing medical healthcare professional (doctor, nurse or HIV counsellor that performs HIV testing with Rapid Tests).
* Any condition which, in the opinion of the Observer, would make the participant unsuitable or unsafe for enrolment or could interfere with the completion of the assessment, consent form and questionnaire etc. or bias the outcome (e.g. being unable to see/read by forgetting to bring reading glasses, being intoxicated, acute sickness, visibly distressed).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-12-10 (Estimated)

PRIMARY OUTCOMES:
Percent positive and negative agreement of the Multiplo® TP/HIV Self-Test to the Participant's HIV and/or syphilis status confirmed by the lab results. | 6 months
  The primary outcome for the study will be the percent positive and negative agreement of the Multiplo® TP/HIV Self-Test to the Participant's HIV and/or syphilis status confirmed by the lab results.
  The percentages for positive and negative agreement will be calculated with the two-sided 95% confidence intervals for both as follows:
  * Positive Agreement= ((n) HIV or syphilis Multiplo reactive results )/((n) HIV or syphilis positive status)×100
  * Negative Agreement= ((n)HIV or syphilis Multiplo non reactive results )/((n) HIV or syphilis negative status)×100 Percent positive and negative agreement will be calculated for each analyte (HIV or syphilis) separately.
Descriptive analysis of sociodemographic characteristics of people experiencing homelessness who are accessing HIV and Syphilis testing | 6 months
  The embedded study aims to understand the sociodemographic and health profile of PEH accessing WHIWH. Descriptive analysis of sociodemographic variables, risk behaviours, HIV/syphilis testing variables will be completed.

SECONDARY OUTCOMES:
Percent of correctly interpreted mock devices by self-test participants. | 6 months
  Participants will answer a series of questions after they complete the Multiplo® TP/HIV Self-Test assessment and Interpretation of Results - Mock Devices. Participants will be given a panel of contrived devices and asked to interpret the results of the contrived devices. Participant answers will be compared to known results from the assigned panels.
Rates of Positive HIV and Syphilis and rates of first time testers among people experiencing homelessness | 6 months
  Number of PEH who have tested positive for HIV and/or syphilis in the laboratory test. Number of PEH tested for HIV and/or syphilis for the first time through the project. Number of PEH who have been tested for HIV and/or syphilis before the intervention and which type of service.

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Cool Aid Community Health Centre, Victoria, British Columbia
  - Hassle Free Clinic, Toronto, Ontario
  - Women's Health in Women's Hands, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] Allen CG, Barbero C, Shantharam S, Moeti R. Is Theory Guiding Our Work? A Scoping Review on the Use of Implementation Theories, Frameworks, and Models to Bring Community Health Workers into Health Care Settings. J Public Health Manag Pract. 2019 Nov/Dec;25(6):571-580. doi: 10.1097/PHH.0000000000000846. PMID 30180116
- [Background] Israel BA, Schulz AJ, Parker EA, Becker AB. Critical Issues in Developing and Following Community-Based Participatory Research Principles. In: Minkler M, Wallerstein N, editors. Community-Based Participatory Research for Health. Jossey-Bass; 2008. p. 47-62.
- [Background] Scott K, Beckham SW, Gross M, Pariyo G, Rao KD, Cometto G, Perry HB. What do we know about community-based health worker programs? A systematic review of existing reviews on community health workers. Hum Resour Health. 2018 Aug 16;16(1):39. doi: 10.1186/s12960-018-0304-x. PMID 30115074
- [Background] Berg RC, Page S, Ogard-Repal A. The effectiveness of peer-support for people living with HIV: A systematic review and meta-analysis. PLoS One. 2021 Jun 17;16(6):e0252623. doi: 10.1371/journal.pone.0252623. eCollection 2021. PMID 34138897
- [Background] Mwai GW, Mburu G, Torpey K, Frost P, Ford N, Seeley J. Role and outcomes of community health workers in HIV care in sub-Saharan Africa: a systematic review. J Int AIDS Soc. 2013 Sep 10;16(1):18586. doi: 10.7448/IAS.16.1.18586. PMID 24029015
- [Background] Jackson C, Tremblay G. Accelerating our response: Government of Canada five-year action plan on sexually transmitted and blood-borne infections. Can Commun Dis Rep. 2019 Dec 5;45(12):323-326. doi: 10.14745/ccdr.v45i12a04. eCollection 2019 Dec 5. PMID 32167085
- [Background] Canadian Institutes of Health Research. CIHR HIV/AIDS and STBBI research initiative strategic plan 2022-2027. Ottawa: Canadian Institutes of Health Research = Instituts de recherche en santé du Canada; 2022.
- See also: The Street Health Report 2007 | The Homeless Hub — https://www.homelesshub.ca/resource/street-health-report-2007
- See also: BC Public Advisory Network. What is Community-Based Research? — https://paninbc.ca/research-and-evaluation/what-is-cbr/
- See also: Canadian Definition of Homelessness | The Homeless Hub — https://www.homelesshub.ca/resource/canadian-definition-homelessness